CLINICAL TRIAL: NCT03286556
Title: Study of Therapeutic Plasma Exchange, Rituximab and Intravenous Immunoglobulin for Acute Exacerbations of Idiopathic Pulmonary Fibrosis (STRIVE-IPF)
Brief Title: Autoantibody Reduction for Acute Exacerbations of Idiopathic Pulmonary Fibrosis
Acronym: STRIVE-IPF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Brigham and Women's Hospital (Other); Temple University (Other); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Steven R. Duncan, MD, Prinicpal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F170530011; 1U01HL133232-01A1 (NIH)
Record Dates: First submitted 2017-09-12; First posted 2017-09-18 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Idiopathic Pulmonary Fibrosis, Acute Fatal Form
Keywords: Acute Exacerbation of Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Therapeutics; Anti-Bacterial Agents; Steroids

STUDY DESIGN:
Intervention Model Description: Open label randomized controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Autoantibody Reductive Therapy (Experimental): Therapeutic Plasma Exchange (TPE) consisting of 1x estimated plasma volume exchanges for 3 successive days (1-3) and then, after a one day interval to enable equilibration of autoantibodies between intra- and extra-vascular spaces, again on days 5, 6, 9, 11, 13, and 15.
  Rituximab: One gm i.v. will be administered on day 6 and day 15 after completion of the TPE on those days.
  Intravenous immunoglobulin (IVIG): 0.5 gm/kg/day i.v. on days 16-19
  All subjects in this trial, including patients in this arm, will receive identical empiric antibiotics and steroids. The steroid dose is: Prednisone 60 mg (p.o.) on day 1, followed by 20 mg/day on days 2-5, 7-14, and 16-19 (or the i.v. methylprednisolone equivalent). Methylprednisolone 100 mg i.v. will be administered on days 6 and 15, as a premedication prior to the rituximab.
  Interventions: Drug: Autoantibody Reductive Therapy
- Treatment as Usual (TAU) (Active Comparator): The same steroid regimen as described for the experimental arm, i.e., prednisone 60 mg (p.o.) on day 1, followed by 20 mg/day on days 2-5, 7-14, and 16-19 (or the i.v. methylprednisolone equivalent), and methylprednisolone 100 mg i.v. administered on days 6 and 15, as well as empiric antibiotics.
  Interventions: Drug: Treatment as Usual (TAU)

INTERVENTIONS:
Drug: Autoantibody Reductive Therapy — TPE x 9, rituximab x 2, IVIG x 4. See arm/group descriptions for additional details.
  Arms: Autoantibody Reductive Therapy
Drug: Treatment as Usual (TAU) — Antibiotics and steroids
  Other Names: Antibiotics and steroids
  Arms: Treatment as Usual (TAU)

SUMMARY:
Acute exacerbations (AE) are a dreaded manifestation of idiopathic pulmonary fibrosis (IPF) that presents with rapidly worsening respiratory function over days to weeks. AE account for about 1/2 the deaths in IPF patients, and are refractory to all medical therapies attempted to date.

Considerable preliminary data shows pathological B-cell abnormalities and autoantibodies are present in AE-IPF and associated with disease severity.

The experimental therapy here (therapeutic plasma exchange plus rituximab plus intravenous immunoglobulin) is mechanistically targeted to ameliorate autoantibody-mediated pulmonary injury. Anecdotal pilot studies indicate these treatments have significant benefit for a disease syndrome that has, until now, been almost invariably inexorable. This clinical trial has the potential to profoundly affect current paradigms and treatment approaches to patients with AE-IPF.

DETAILED DESCRIPTION:
The primary goal of clinical trial is to determine effects of combined therapeutic plasma exchange (TPE), rituximab, and intravenous immunoglobulin (IVIG) in comparison to effects of treatment as usual (TAU), among AE-IPF patients.

Our central hypothesis is "AUTOANTIBODY REDUCTION IS BENEFICIAL FOR AE-IPF PATIENTS." A corollary of this hypothesis is that antibody-mediated autoimmunity can play an important role in IPF exacerbations.

Following baseline screening assessments, hospitalized AE-IPF patients at the collaborating sites that meet all inclusion/exclusion criteria will be randomly assigned to receive one of the following treatments in a ratio of 2:1:

• Arm A (n=34) - Experimental Treatment:

Steroids: Prednisone 60 mg (p.o.) on day 1, followed by 20 mg/day on days 2-5, 7-14, and 16-19 (or the i.v. methylprednisolone equivalent). Methyl-prednisolone 100 mg i.v. will be administered on days 6 and 15, as a premedication prior to the rituximab.

Insertion of a dialysis/apheresis catheter into a central vein, and initiation of therapeutic plasma exchange (TPE), rituximab, and intravenous immunoglobulin (IVIG) regimens:

Therapeutic Plasma Exchange (TPE) will consist of 1x estimated plasma volume exchanges for 3 successive days (1-3) and then, after a one day interval to enable equilibration of autoantibodies between intra- and extra-vascular spaces, again on days 5, 6, 9, 11, 13, and 15.

Rituximab: One gm i.v. will be administered on day 6 and day 15 after completion of the TPE on those days.

Intravenous immunoglobulin (IVIG): 0.5 gm/kg/day i.v. on days 16-19

• Arm B (n=17) - Treatment as Usual (TAU):

The same steroid regimen as described for Arm A, i.e., prednisone 60 mg (p.o.) on day 1, followed by 20 mg/day on days 2-5, 7-14, and 16-19 (or the i.v. methylprednisolone equivalent), and methylprednisolone 100 mg i.v. administered on days 6 and 15.

All patients enrolled in both cohorts at all sites will also receive empiric broad-spectrum antibiotics for 8 days. The empiric antibiotic regimen will be reassessed and tailored based on any subsequent cultures and sensitivity results.

Patients will be monitored carefully for occurrences of adverse events, laboratory test abnormalities, and changes in vital signs.

The respective treatment courses can be finished on an outpatient basis among enrolled patients who are able to be discharged from the hospital, if medically indicated, and if those treatment compliance can be assured.

Patients will be followed for the duration of their hospital admission after enrollment, and then observed as either inpatients or outpatients on days 19, 60, 90, 180, 270, and 365. A telephone contact will occur at monthly intervals, aside from those visits above. The total observation/subject is 365 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40-85 years old.
2. A diagnosis of IPF that fulfills ATS/ERS Consensus Criteria.1
3. Worsening or new development of dyspnea or hypoxemia within the last 30 days.
4. Ground-glass abnormality and/or consolidation superimposed on a reticular or honeycomb usual interstitial pneumonitis (UIP) pattern on locally read chest CT scan.
5. Ability and willingness to give informed consent (no surrogates) and adhere to study requirements.

Exclusion Criteria:

1. Diagnoses of current infection per clinical or microbial assessments.
2. Diagnoses of an additional or alternative etiology for respiratory dysfunction based upon clinical assessment, including congestive heart failure, sepsis, thromboembolism, etc.
3. History or serologic evidence of hepatitis B or C infection.
4. Coagulopathy, defined as a International Normalized Ratio (INR) >1.6, partial thromboplastin time (PTT) > 2x control, fibrinogen <100 mg/dL, or platelet count <50 thousand (K) unless these abnormalities can be reversed safely.
5. Hyperosmolar state or diabetic ketoacidosis to suggest uncontrolled diabetes, or uncontrolled hypertension (systolic BP >160 mm Hg and diastolic BP >100 mm Hg) that would contraindicate use of corticosteroids.
6. Hemodynamic instability, defined as an inotrope or vasopressor requirement.
7. History of reaction to blood products or murine-derived products or prior rituximab use.
8. History of malignancy, excluding basal or squamous cell skin cancer and low-risk prostate cancer, the latter defined as stage T1 or T2a, with prostate specific antigen (PSA) less than 10 ng/dl. The experimental treatments are not known to promote cancer progression, and these criteria are within current guidelines.
9. Unwillingness to accept blood product transfusion.
10. Diagnosis of major comorbidities expected to interfere with study participation.
11. Treatment for >14 days within the preceding month with >20 mg. prednisone (or equivalent) or any treatment during the last month with a cellular immuno-suppressant (e.g., cyclophosphamide, methotrexate, calcineurin inhibitors, mycophenolate, azathioprine, etc.). An exception will be made if the patient has a bronchoalveolar lavage (BAL) negative for pathogens.
12. Current treatment with an angiotensin converting enzyme inhibitor that cannot be discontinued and/or substituted (to obviate hemodynamic complications during TPE).
13. Concurrent participation in other experimental trials.
14. Fertile females who do not agree to contraception or abstinence, or have a positive pregnancy test (urine or blood). IPF is a disease of older adults, and male predominant, so this will not be a frequent consideration.
15. Presence of positive (abnormal) classical autoimmune tests: anti-nuclear antibody (ANA), rheumatoid factor (RF), Anti- Sjögren's-syndrome-related antigen (SSA) , and Anti-Cyclic Citrullinated Peptide (CCP). This criterion will eliminate patients with confounding classical autoimmune syndromes. Many IPF patients will have already had these tests, which are standard of practice (SOP) at many IPF centers, and these prior results will suffice if the tests were performed within the last year. Otherwise, these tests need to be performed prior to enrollment and they can usually be procured in 1-2 days. Based on experience, we anticipate ~10% of patients who fulfill all other IPF criteria will nonetheless be positive for one of these classical autoantibody tests.
16. IgA deficiency (IgA level <7 mg/dL)- to preclude IVIG reactions.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Survival | 6 months
  Actuarial survival

SECONDARY OUTCOMES:
Oxygen requirements | 6 months
  Measures of oxygen required to maintain arterial oxygen concentration (SaO2) >/=93%
Walk distance | 6 months
  6 minute walk distance using standardized American Thoracic Society/European Respiratory Society (ATS/ERS) protocols.
Adverse Events | Through study completion, an average of 1 year
  The presence of adverse events attributable to the trial intervention

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Dan Dilling, Chicago, Illinois
  - Thomas Jefferson University Medical Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor University Medical Center, Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Feghali-Bostwick CA, Tsai CG, Valentine VG, Kantrow S, Stoner MW, Pilewski JM, Gadgil A, George MP, Gibson KF, Choi AM, Kaminski N, Zhang Y, Duncan SR. Cellular and humoral autoreactivity in idiopathic pulmonary fibrosis. J Immunol. 2007 Aug 15;179(4):2592-9. doi: 10.4049/jimmunol.179.4.2592. PMID 17675522
- [Result] Gilani SR, Vuga LJ, Lindell KO, Gibson KF, Xue J, Kaminski N, Valentine VG, Lindsay EK, George MP, Steele C, Duncan SR. CD28 down-regulation on circulating CD4 T-cells is associated with poor prognoses of patients with idiopathic pulmonary fibrosis. PLoS One. 2010 Jan 29;5(1):e8959. doi: 10.1371/journal.pone.0008959. PMID 20126467
- [Result] Xue J, Gochuico BR, Alawad AS, Feghali-Bostwick CA, Noth I, Nathan SD, Rosen GD, Rosas IO, Dacic S, Ocak I, Fuhrman CR, Cuenco KT, Smith MA, Jacobs SS, Zeevi A, Morel PA, Pilewski JM, Valentine VG, Gibson KF, Kaminski N, Sciurba FC, Zhang Y, Duncan SR. The HLA class II Allele DRB1*1501 is over-represented in patients with idiopathic pulmonary fibrosis. PLoS One. 2011 Feb 23;6(2):e14715. doi: 10.1371/journal.pone.0014715. PMID 21373184
- [Result] Kahloon RA, Xue J, Bhargava A, Csizmadia E, Otterbein L, Kass DJ, Bon J, Soejima M, Levesque MC, Lindell KO, Gibson KF, Kaminski N, Banga G, Oddis CV, Pilewski JM, Sciurba FC, Donahoe M, Zhang Y, Duncan SR. Patients with idiopathic pulmonary fibrosis with antibodies to heat shock protein 70 have poor prognoses. Am J Respir Crit Care Med. 2013 Apr 1;187(7):768-75. doi: 10.1164/rccm.201203-0506OC. PMID 23262513
- [Result] Xue J, Kass DJ, Bon J, Vuga L, Tan J, Csizmadia E, Otterbein L, Soejima M, Levesque MC, Gibson KF, Kaminski N, Pilewski JM, Donahoe M, Sciurba FC, Duncan SR. Plasma B lymphocyte stimulator and B cell differentiation in idiopathic pulmonary fibrosis patients. J Immunol. 2013 Sep 1;191(5):2089-95. doi: 10.4049/jimmunol.1203476. Epub 2013 Jul 19. PMID 23872052
- [Result] Vuga LJ, Tedrow JR, Pandit KV, Tan J, Kass DJ, Xue J, Chandra D, Leader JK, Gibson KF, Kaminski N, Sciurba FC, Duncan SR. C-X-C motif chemokine 13 (CXCL13) is a prognostic biomarker of idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2014 Apr 15;189(8):966-74. doi: 10.1164/rccm.201309-1592OC. PMID 24628285
- [Result] Donahoe M, Valentine VG, Chien N, Gibson KF, Raval JS, Saul M, Xue J, Zhang Y, Duncan SR. Autoantibody-Targeted Treatments for Acute Exacerbations of Idiopathic Pulmonary Fibrosis. PLoS One. 2015 Jun 17;10(6):e0127771. doi: 10.1371/journal.pone.0127771. eCollection 2015. PMID 26083430
- [Result] Collard HR, Moore BB, Flaherty KR, Brown KK, Kaner RJ, King TE Jr, Lasky JA, Loyd JE, Noth I, Olman MA, Raghu G, Roman J, Ryu JH, Zisman DA, Hunninghake GW, Colby TV, Egan JJ, Hansell DM, Johkoh T, Kaminski N, Kim DS, Kondoh Y, Lynch DA, Muller-Quernheim J, Myers JL, Nicholson AG, Selman M, Toews GB, Wells AU, Martinez FJ; Idiopathic Pulmonary Fibrosis Clinical Research Network Investigators. Acute exacerbations of idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2007 Oct 1;176(7):636-43. doi: 10.1164/rccm.200703-463PP. Epub 2007 Jun 21. PMID 17585107
- [Derived] Kulkarni T, Criner GJ, Kass DJ, Rosas IO, Scholand MB, Dilling DF, Summer R, Duncan SR. Design of the STRIVE-IPF trial- study of therapeutic plasma exchange, rituximab, and intravenous immunoglobulin for acute exacerbations of idiopathic pulmonary fibrosis. BMC Pulm Med. 2024 Mar 20;24(1):143. doi: 10.1186/s12890-024-02957-3. PMID 38509495
- [Derived] Kulkarni T, Criner GJ, Kass DJ, Rosas IO, Scholand MB, Dilling DF, Summer R, Duncan SR. Design of the STRIVE-IPF Trial- Study of Therapeutic Plasma Exchange, Rituximab, and Intravenous Immunoglobulin for Acute Exacerbations of Idiopathic Pulmonary Fibrosis. Res Sq [Preprint]. 2024 Feb 28:rs.3.rs-3962419. doi: 10.21203/rs.3.rs-3962419/v1. PMID 38464052